CLINICAL TRIAL: NCT03443323
Title: Evaluation of Organizational Skills Training (OST) Program for Upper Elementary Students
Brief Title: Organizational Skills Training - Tier 2 (OST-T2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); New York University (Other); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-014227; R305A170052-20 (Other Grant/Funding Number: US Dept. of Education)
Record Dates: First submitted 2017-11-28; First posted 2018-02-23 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Executive Function; Behavioral Research; Schools; Behavior Therapy
Keywords: Executive Function; Behavioral Research; Cost Analysis; Students; Schools; Randomized Controlled Trial; Behavior Therapy; Skills Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OST-T2 Intervention group (Experimental): Small group skills training for students in grades 3 through 5 with difficulties with organization, time management, and planning skills. Includes parent and teacher involvement to support student skills use.
  Interventions: Behavioral: Organizational Skills Training - Tier 2 (OST-T2)
- Treatment as usual control group (No Intervention): Strategies currently in use by schools to address organization, time management, and planning skills problems.

INTERVENTIONS:
Behavioral: Organizational Skills Training - Tier 2 (OST-T2) — OST-T2 is a small group skills training intervention, with parents and teachers supporting children's use of new skills. The program manual includes strategies for training and coaching school staff, referred to as school partners, to effectively implement OST-T2 and guidelines to modify the program for implementation in diverse schools with diverse students. Each student session includes: (a) homework review to assess completion of between-session skills implementation; (b) skill-building activities, which include the use of modeling, shaping, guided practice, and reinforcement for organized behavior; and (c) activities to promote generalization of skills. Sessions address four organizational challenges: (a) tracking assignments, (b) managing materials, (c) managing time, and (d) planning for long term assignments.
  Arms: OST-T2 Intervention group

SUMMARY:
The purpose of this study was to evaluate the Organizational Skills Training Program - Tier 2 version (OST-T2) in a cluster randomized trial. Participating schools will be randomly assigned to one of two groups: 1) an OST-T2 intervention group and 2) a treatment as usual control group. Participating students (3rd through 5th grade) were from 22 schools in Pennsylvania and New Jersey and included both urban and suburban schools serving a diverse population. OST-T2 is a small-group, skills training intervention for children, which includes parent and teacher consultation to support student use of new skills. The program is delivered by school staff who receive training and consultation from intervention experts.

DETAILED DESCRIPTION:
Context: Although multiple factors influence school functioning, executive function (EF) deficits have been found to be a key predictor of academic achievement. EF is a higher order cognitive ability associated with persistent goal-directed behavior. Organization, time management, and planning (OTMP) skills are aspects of EF that are particularly associated with children's academic performance. Organizational demands increase over the course of early schooling and are relatively high by 3rd through 5th grade. Poor OTMP skills during this period adversely impact academic functioning. In the late elementary school grades, as students are expected to become more organized, some students have difficulty learning these skills in spite of classroom supports provided by teachers, placing them at increased risk for academic failure.

Objectives: The purpose of this study was to conduct an evaluation of the Organizational Skills Training Program - Tier 2 version (OST-T2), a fully developed intervention for students in general education. The proposed study builds upon research demonstrating the efficacy of a clinic-based version of the OST intervention (OST-C) in remediating OTMP skills deficits and improving academic functioning for 3rd, 4th and 5th graders with attention-deficit hyperactivity disorder (ADHD), and a recent pilot research demonstrating the feasibility and potential effectiveness of a school-based version of OST provided by end users ("school partners") for 3rd through 5th graders. It also builds upon research training school staff to implement evidence-based interventions with high fidelity.

Study Design: This is a cluster-randomized trial with a treatment as usual (TAU) control group.

Setting/Participants: Schools (22) were located in Pennsylvania and New Jersey and include urban and suburban schools serving a diverse population. Students (3rd to 5th grade) who are struggling the most with OTMP deficits and whose academic performance is negatively impacted by their OTMP deficits will be referred to the study team by their general education teachers.

Study Interventions and Measures: OST-T2 is a small group skills training intervention, with parents and teachers supporting children's use of new skills. The program manual includes strategies for training and coaching school staff, referred to as school partners, to effectively implement OST-T2 and guidelines to modify the program for implementation in diverse schools with diverse students. Each student session includes: (a) homework review to assess completion of between-session skills implementation; (b) skill-building activities, which include the use of modeling, shaping, guided practice, and reinforcement for organized behavior; and (c) activities to promote generalization of skills. Sessions address four organizational challenges: (a) tracking assignments, (b) managing materials, (c) managing time, and (d) planning for long term assignments.

Investigators measured the following: intervention fidelity, stakeholder engagement, student OTMP skills, student academic self-efficacy, student academic outcomes, student characteristics, feasibility, usability, and acceptability of OST-T2. In addition, investigators tracked the interventions that are offered as treatment-as-usual in TAU schools. A cost analysis related to the implementation of OST-T2 will also be completed.

ELIGIBILITY:
Inclusion Criteria:

Any student enrolled in grades 3 through 5 in one of the participating schools who meets the following criteria.

1. First, students will be recommended by their general education teacher if the following are true: (a) students who are struggling the most with OTMP skills, (b) whose OTMP skill deficits are the students' primary concern (c) whose academic performance is negatively impacted by their OTMP deficits, and (d) who have at least one parent who speaks English.
2. Second, students must have or be at risk for developing OTMP deficits.

Exclusion Criteria:

1. Students will be excluded if they are in a pull-out special education classroom for more than 50% of the day as the organizational demands for these students may differ from those students placed mostly in general education.
2. Students with a one-to-one aide will be excluded because the presence of an aide substantially alters how an organizational intervention is implemented.
3. Students from families in which both caregivers do not speak English will be excluded because the program has not yet been developed for non-English speakers.
4. Only one student per family will be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Power, PhD, Principal Investigator — Children's Hospital of Philadelphia; Jenelle Nissley-Tsiopoinis, PhD, Principal Investigator — Children's Hospital of Philadelphia; Jennifer Mautone, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - New York University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Per Institute for Educational Sciences (IES) requirements, the timeframe for accessibility of data will be reviewed during each annual progress review and revised as necessary. The final dataset will be exported from REDCap to Microsoft Excel and commonly used statistical software packages such as SPSS and SAS, as requested by the individuals seeking access to the data. The research team will prepare a codebook to share with the requesting individuals. The codebook will provide information about all of the variables and how the composite variables (e.g. factor scores) were derived.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become accessible after the study is completed and primary study findings are published in a peer-reviewed journal. Data will be available for 10 years from that time. Per Institute for Educational Sciences (IES) requirements, the timeframe for accessibility of data will be reviewed during each annual progress review and revised as necessary.
Access Criteria: Individuals interested in using the data should contact Dr. Thomas Power (power@chop.edu). When our research team receives a request for access to the data a data file and supporting documentation will be prepared by the research team. Only de-identified data will be made accessible in order to prevent identification of students, parents, and school staff who participated in this project. Per Children's Hospital of Philadelphia (CHOP) policies, a data use agreement is necessary prior to sharing data.

REFERENCES:
- [Background] Best JR, Miller PH, Naglieri JA. Relations between Executive Function and Academic Achievement from Ages 5 to 17 in a Large, Representative National Sample. Learn Individ Differ. 2011 Aug;21(4):327-336. doi: 10.1016/j.lindif.2011.01.007. PMID 21845021
- [Background] Best JR, Miller PH, Jones LL. Executive Functions after Age 5: Changes and Correlates. Dev Rev. 2009 Sep 1;29(3):180-200. doi: 10.1016/j.dr.2009.05.002. PMID 20161467
- [Background] Abikoff, H., & Gallagher, R. (2009). Children's organizational skills scales (COSS), technical manual. North Tonawanda, NY: Multi-Health Systems.
- [Background] Abikoff H, Gallagher R, Wells KC, Murray DW, Huang L, Lu F, Petkova E. Remediating organizational functioning in children with ADHD: immediate and long-term effects from a randomized controlled trial. J Consult Clin Psychol. 2013 Feb;81(1):113-28. doi: 10.1037/a0029648. Epub 2012 Aug 13. PMID 22889336
- [Background] Eiraldi R, McCurdy B, Khanna M, Mautone J, Jawad AF, Power T, Cidav Z, Cacia J, Sugai G. A cluster randomized trial to evaluate external support for the implementation of positive behavioral interventions and supports by school personnel. Implement Sci. 2014 Jan 15;9:12. doi: 10.1186/1748-5908-9-12. PMID 24428904
- [Background] Langberg JM, Dvorsky MR, Evans SW. What specific facets of executive function are associated with academic functioning in youth with attention-deficit/hyperactivity disorder? J Abnorm Child Psychol. 2013 Oct;41(7):1145-59. doi: 10.1007/s10802-013-9750-z. PMID 23640285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Nov., 2017 through Jan., 2022 from 22 schools serving students in upper elementary school in the Philadelphia, PA region.
Pre-assignment Details: Data from 186 student participants were evaluated for this study. Data were derived from parents, teachers, and child self-report. One participant of the 186 was withdrawn prior to the intervention period because this student was found not to meet study eligibility criteria.
Units Other Than Participants: Schools
Groups:
- Treatment as Usual Wait List Control Group: Students in the treatment as usual wait list control group have access to any services and supports their school typically provides to address organization, time management, and planning difficulties. This group receives the OST-T2 intervention after collection of the 12-month follow up data.
Period: Overall Study
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Started | 98; 12 Schools | 88; 10 Schools
Baseline Data (Data pertaining to participating students were collected at all time points from parents, teachers, and students.) | 96; 12 Schools | 88; 10 Schools
Completed (Post-treatment (14 weeks)) | 95; 12 Schools | 86; 10 Schools
Not Completed | 3; 0 Schools | 2; 0 Schools
Not completed — Lost to Follow-up | 2 | 2
Not completed — PI withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Population: The PIs withdrew one participant before the study intervention period because this person was found not to meet study eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Control Group | Total
Number analyzed (Participants) | 97 | 88 | 185
Age, Continuous [Mean (Standard Deviation); unit: Child Age in Years] | 9.8 (0.89) | 9.5 (0.86) | 9.7 (0.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 66 | 56 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 23
  Not Hispanic or Latino | 87 | 75 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 23 | 48
  White | 50 | 55 | 105
  More than one race | 11 | 8 | 19
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 97 | 88 | 185
Child Grade in School [Count of Participants; unit: Participants]
  Grade 3 | 27 | 37 | 64
  Grade 4 | 46 | 32 | 78
  Grade 5 | 24 | 19 | 43
Caregiver mean level of education [Count of Participants; unit: Participants]
  High School Graduate or Less | 13 | 22 | 35
  Partial College/Specialized Training | 30 | 36 | 66
  Standard College or Graduate Degree | 51 | 30 | 81
Family Neighborhood Area Deprivation Index, National Percentile [Mean (Standard Deviation); unit: Percentile] | 39.3 (24.1) | 52.8 (23.8) | 45.7 (24.8)
Child Attention Problems (Behavior Assessment Scale for Children, Third Edition; BASC-3) [Mean (Standard Deviation); unit: T-score] — Raw scores were converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate higher levels of symptoms/problems. A T-score of 60 refers to a mild elevation in symptoms, a T-score of 65 refers to moderate, and a T-score of 70 refers to high elevation.
  T-score | 61.2 (8.4) | 65.1 (7.4) | 63.0 (8.1)
Child Anxiety (Behavioral Assessment System for Children - Third Edition; BASC-3 [Mean (Standard Deviation); unit: T-Score] — Raw scores were converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate higher levels of symptoms/problems. A T-score of 60 refers to a mild elevation in symptoms, a T-score of 65 refers to moderate, and a T-score of 70 refers to high elevation.
  T-Score | 54.1 (11.8) | 53.7 (9.7) | 53.9 (10.8)
Child Autism Spectrum Rating Scale [Mean (Standard Deviation); unit: T-Score] — Raw scores were converted to T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate higher levels of symptoms/problems. A T-score of 60 refers to a mild elevation in symptoms, a T-score of 65 refers to moderate, and a T-score of 70 refers to high elevation.
  T-Score | 50.9 (10.8) | 54.1 (8.3) | 52.5 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Students' Organizational Functioning - Teacher Report
Description: The Children's Organizational Skills Scales - Teacher Version (COSS-T) was used to assess changes in OTMP functioning at home and school over several time points. COSS total scores have good discriminant validity and are sensitive to treatment effects. Each COSS version uses a 4-point rating scale (1=Hardly ever or never to 4=Just about all of the time). Higher scores indicate a worse outcome. Although the COSS yields three subscale scores, only the total score of 28 items was used to reduce the number of measures in the analyses. The mean item score was calculated and used in analyses; possible range is from 1 to 4.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 180 participants provided data that were analyzed. Data were missing for 5 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 95 | 85
scores on a scale
  Baseline | 2.89 [2.80 to 2.99] | 2.86 [2.73 to 2.98]
  Post-treatment (14 weeks) | 2.27 [2.12 to 2.41] | 2.71 [2.61 to 2.82]
  5-month follow-up (22 weeks) | 2.32 [2.19 to 2.45] | 2.71 [2.62 to 2.80]
  12-month follow-up (55 weeks) | 2.40 [2.22 to 2.59] | 2.57 [2.45 to 2.70]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p < .001, Mixed Models Analysis — Statistical significance was evaluated using a threshold p value of .0083, accounting for the estimation of three contrasts of time-by-treatment differences per outcome and two measures per domain (OTMP skills [COSS-P, COSS-T])

2. Primary Outcome: Students' Organizational Functioning - Parent Report
Description: The Children's Organizational Skills Scales - Parent Version (COSS-P) was used to assess changes in OTMP functioning at home and school over several time points. COSS total scores have good discriminant validity and are sensitive to treatment effects. Each COSS version uses a 4-point rating scale (1=Hardly ever or never to 4=Just about all of the time). Higher scores indicate a worse outcome. Although the COSS yields three subscale scores, only the 26-item total score was used to reduce the number of measures in the analyses. The mean item score was calculated and used in analyses; possible range is from 1 to 4.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 183 participants provided data that were analyzed. Data were missing for 2 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 95 | 88
scores on a scale
  Baseline | 2.65 [2.59 to 2.72] | 2.59 [2.53 to 2.64]
  Post-Treatment (14 weeks) | 2.20 [2.09 to 2.31] | 2.51 [2.40 to 2.61]
  5-month follow-up (22 weeks) | 2.25 [2.14 to 2.36] | 2.53 [2.44 to 2.62]
  12-month follow-up (55 weeks) | 2.33 [2.17 to 2.49] | 2.35 [2.18 to 2.51]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Students' Homework Performance - Teacher Report
Description: The Homework Performance Questionnaire (HPQ-T)-Teacher version was used to assess changes in students' homework behavior during the past 4 weeks. Each item is rated on a five-point scale corresponding to amount of time student demonstrated the behavior in the previous 4-week period (0 = 0% to 39% of the time; 1 = 40% to 69% of the time; 2 = 70% to 79% of the time; 3 = 80% to 89% of the time; 4 = 90% to 100% of the time).Higher scores indicate better outcome. The 9-item Student Self-Regulation factor was used in the analyses. This factor has been demonstrated to have strong psychometric properties. Mean item score was used in analyses; possible range is from 0 to 4.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 179 participants provided data that were analyzed. Data were missing for 6 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 95 | 84
scores on a scale
  Baseline | 1.76 [1.38 to 2.14] | 2.07 [1.64 to 2.51]
  Post-treatment (14-weeks) | 2.68 [2.23 to 3.13] | 2.32 [2.12 to 2.53]
  5-month follow-up (22 weeks) | 2.55 [2.17 to 2.93] | 2.44 [2.22 to 2.66]
  12-month follow-up (55 weeks) | 1.97 [1.35 to 2.59] | 2.14 [1.69 to 2.60]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p = 0.007, Mixed Models Analysis — Statistical significance was evaluated using a threshold p value of .0083, accounting for the estimation of three contrasts of time-by-treatment differences per outcome and two measures per domain (homework performance [HPC, HPQ-T])

4. Secondary Outcome: Students' Homework Performance - Parent Report
Description: The Homework Problem Checklist (HPC) is a 20-item parent-report measure that was used to assess changes in student homework performance. Parents indicate the frequency with which student engage in behavior during homework time at home on a four-point scale (0 = never to 3 = very often). The psychometric properties of this instrument have been shown to be acceptable, and the HPC was sensitive to treatment effects in the previous OST-C study. The total HPC score was used in the analyses. Higher scores indicate worse outcomes. Mean item score was calculated and used in analyses; possible range is from 0 to 3.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 183 participants provided data that were analyzed. Data were missing for 2 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 95 | 88
scores on a scale
  Baseline | 1.49 [1.35 to 1.63] | 1.35 [1.23 to 1.47]
  Post-treatment (14 weeks) | 0.94 [0.75 to 1.14] | 1.20 [1.06 to 1.35]
  5-month follow-up (22 weeks) | 0.97 [0.81 to 1.12] | 1.26 [1.11 to 1.41]
  12-month follow-up (55 weeks) | 1.13 [0.95 to 1.32] | 1.14 [0.95 to 1.34]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p < .001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Student Academic Proficiency
Description: The Academic Proficiency Scale (APS) is a teacher-report measure that assesses (changes in) proficiency in six academic subjects relative to standard expectations (1=Well below standard expected at this time of year; 3=At standard; 5=Well above standard). Higher scores indicate a better outcome. Ratings were averaged across six academic subjects; mean item score is the unit of analysis. Possible range is from 1 to 5. Reliability is acceptable (alpha = .84), and this measure is sensitive to OST treatment effects.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 180 participants provided data that were analyzed. Data were missing for 5 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 95 | 85
scores on a scale
  Baseline | 2.59 [2.44 to 2.74] | 2.57 [2.30 to 2.84]
  Post-treatment (14 weeks) | 2.77 [2.60 to 2.94] | 2.54 [2.40 to 2.67]
  5-month follow-up (22 weeks) | 2.80 [2.65 to 2.95] | 2.53 [2.44 to 2.63]
  12-month follow-up (55 weeks) | 2.67 [2.46 to 2.88] | 2.62 [2.34 to 2.90]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p < .06, Mixed Models Analysis — Statistical significance was evaluated using a threshold p value of .0083, accounting for the estimation of three contrasts of time-by-treatment differences per outcome and two measures per domain (academic performance [ACES, APS])

6. Secondary Outcome: Student Academic Competence
Description: The Academic Competence Evaluation Scales (ACES) is a teacher-report scale that assesses changes in the academic competence of students in kindergarten through grade 12. The Reading/Language Arts and Math subscales of this measure were used. Items are rated from 1 = far below to 5 = far above grade level. Higher scores indicate better outcome. Alpha coefficients and test-retest correlations for these subscales have been shown to be above .90. The average item score for Reading/Language Arts (11 items) and Math (8 items) subscales were calculated. Then the average of these subscale scores was used in the analyses. Possible range is from 1 to 5.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 169 participants provided data that were analyzed. Data were missing for 16 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 88 | 81
scores on a scale
  Baseline | 2.46 [2.31 to 2.62] | 2.31 [2.11 to 2.51]
  Post-treatment (14 weeks) | 2.71 [2.55 to 2.88] | 2.35 [2.17 to 2.53]
  5-month follow-up (22 weeks) | 2.72 [2.57 to 2.87] | 2.46 [2.30 to 2.61]
  12-month follow-up (55 weeks) | 2.63 [2.42 to 2.84] | 2.42 [2.20 to 2.63]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p > .0083, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Student Academic Grades
Description: Student report card grades for the first marking period of the year students participate in OST-T2/TAU and for the last marking period of the academic year of participation were used to examine impact on academic performance. Grades were harmonized across participating school districts to a uniform grading scale (ranging from low of 1 to high of 4). A composite academic grade score was computed for each student based on their grades in math and reading/language arts (possible range = 1 to 4). Higher scores indicate better outcomes.
Time Frame: Baseline, 5-months
Population: Note that 165 participants provided data that were analyzed. Data were missing for 20 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 89 | 76
scores on a scale
  Baseline | 2.50 [2.29 to 2.69] | 2.52 [2.32 to 2.72]
  5-month follow-up (22 weeks) | 2.72 [2.49 to 2.94] | 2.71 [2.52 to 2.91]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p > .05, Mixed Models Analysis — Statistical significance was evaluated using a threshold p value of .05

8. Secondary Outcome: Student Self-efficacy
Description: Patterns of Adaptive Learning Scales (PALS) was used to evaluate changes in students' perceptions of their ability to overcome challenges to perform their class work (e.g., "I can do even the hardest work in this class if I try."). Items are rated on a 5-item scale from 1 = not at all true to 5 = very true. Higher scores indicate better outcomes. Mean item scores were used in analyses; possible range is from 1 to 5.
Time Frame: Baseline, 14-weeks (post-treatment), 5-months and 12-months
Population: Note that 181 participants provided data that were analyzed. Data were missing for 4 participants on this measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Wait List Control Group
Number analyzed (Participants) | 97 | 84
scores on a scale
  Baseline | 3.90 [3.69 to 4.10] | 3.88 [3.78 to 3.97]
  Post-treatment (14 weeks) | 4.09 [3.89 to 4.29] | 3.98 [3.87 to 4.10]
  5-month follow-up (22 weeks) | 4.18 [4.03 to 4.34] | 4.08 [3.84 to 4.31]
  12-month follow-up (55 weeks) | 4.12 [3.75 to 4.48] | 4.22 [3.87 to 4.57]
Statistical Analysis 1: Comparison: OST-T2 Intervention Group vs Treatment as Usual Wait List Control Group; Test type: Superiority; p > .05, Mixed Models Analysis — Statistical significance was evaluated using a threshold p value of .05

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | OST-T2 Intervention Group | Treatment as Usual Control Group
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/88
Other Adverse Events (participants affected / at risk) | 0/97 | 0/88

LIMITATIONS AND CAVEATS:
Findings are generalizable to schools for which OST-T2 was viewed as aligned with school mission, feasible to deliver, and could be implemented by a school professional. Children identified as Black or White were overrepresented; those identified as Hispanic/Latino were underrepresented. Schools serving a high proportion of children living in poverty/deep poverty were underrepresented. COVID-19 resulted in participation challenges that limited the final sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03443323/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03443323/SAP_001.pdf
  • Informed Consent Form (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03443323/ICF_002.pdf